CLINICAL TRIAL: NCT02504047
Title: Use of Haploidentical Related Donors for Patients Without Matched Sibling, Unrelated Donor or Cord Blood Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: The Canadian Blood and Marrow Transplant Group (Network)
Responsible Party: Principal Investigator, Andrew Daly, MD, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26110
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hematologic Neoplasms
Keywords: Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T-Cell replete haplo-transplant (Experimental): Infusion of peripheral blood stem cells from a haploidentical related donor following myeloablative conditioning. Cyclophosphamide, mycophenolate mofetil and tacrolimus will be given for GVHD prophylaxis.
  Interventions: Procedure: T-Cell replete haplo-transplant

INTERVENTIONS:
Procedure: T-Cell replete haplo-transplant — Infusion of haploidentical related donor peripheral blood stem cells following myeloablative conditioning (fludarabine 200 mg/m2, busulfan 12.8 mg/kg and total body irradiation (TBI) 400 centigray -or- fludarabine 200 mg/m2, busulfan 9.6 mg/kg). GVHD prophylaxis will be with cyclophosphamide 50 mg/kg/day x 2 on days 3 & 4, mycophenolate mofetil 1 gm p.o. bid days 5 - 35 and tacrolimus (5-15 ug/ml) days 5 - 100.

SUMMARY:
The administration of high-dose chemotherapy followed by the infusion of blood or bone marrow stem cells (stem cell transplantation) from a matched donor has become standard treatment for patients with high-risk or relapsed hematological cancers. Currently, donors are found for approximately 80% of people who require such treatment, although the chance of finding a donor is much lower in some ethnic communities. In the current study the investigators will offer patients requiring transplantation, but for whom well matched donors cannot be identified either from within the family or on the donor registry, a transplant from a half-matched (haploidentical) family member. A myeloablative conditioning regimen and un-manipulated peripheral blood stem cells will be used. Post-transplant cyclophosphamide, tacrolimus and mycophenolate mofetil will be used to prevent graft versus host disease (GVHD). The primary outcome measure will be 6 month survival free from graft failure, relapse and grade 3-4 acute GVHD. Other outcomes of interest will include the frequency of Cytomegalovirus (CMV) or Epstein-Barr Virus (EBV) requiring treatment, overall survival and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* A hematological malignancy such as acute leukemia or myelodysplastic syndrome requiring hematopoietic stem cell transplantation.
* A haploidentical family member willing to donate.
* Suitable performance status, organ function (as defined locally) and disease status for transplantation.
* Patients with acute leukemia must be in morphological complete remission. Patients with chronic myelogenous leukemia must be in chronic phase and those with lymphoma must have chemosensitive disease (at least partial remission to most recent chemotherapy regimen).
* Given written, informed consent to participate in a clinical trial.

Exclusion Criteria:

* An 8/8 matched sibling donor or matched unrelated donor (based on high-resolution typing as appropriate), available within a time frame acceptable to the treating physician
* Patients with an available single allele or single antigen mismatched donor (7/8 or 9/10) or available cord blood donor can be included at the discretion of the treating team, according to local institutional practice.
* Prior allogeneic transplant
* Any exclusion criteria for allogeneic stem cell transplant, as defined by the program. Examples typically include pregnancy, significant comorbidity, and active uncontrolled infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Six month survival, free from relapse, graft failure and grade III/IV acute GVHD | Six months

SECONDARY OUTCOMES:
Incidence of Grade III/IV Acute Graft Versus Host Disease | Six months
Incidence of Chronic Extensive Graft Versus Host Disease | One year
Cumulative incidence of non-relapse mortality at 1 year | One year
Graft failure rate (ANC < 0.5 and low donor chimerism) | Six months
Overall and Disease Free Survival | One year
Relapse Rate | One year
Patients remaining on immune suppression at 1 year | One year
Incidence of CMV and EBV reactivation requiring treatment | One year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Daly, MD, Principal Investigator — University of Calgary; Kristjan Paulson, MD, Principal Investigator — University of Manitoba
Locations (5):
- Canada (5):
  - Foothills Medical Center / Tom Baker Cancer Center, Calgary, Alberta
  - Health Sciences Center, Winnipeg, Manitoba
  - Ottawa General Hospital, Ottawa, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan